CLINICAL TRIAL: NCT00541723
Title: A Prospective, Randomized, Double-Blind, Multicenter Trial to Investigate the Efficacy and Safety of NT 201 in Comparison to Placebo and to Compare Two Different Application Schemes of NT 201 in the Treatment of Lateral Periorbital Wrinkles
Brief Title: Efficacy and Safety of NT 201 in the Treatment of Lateral Periorbital Wrinkles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRZ 60201-0617/1; 2006-005396-17 (EudraCT Number)
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Lateral Periorbital Wrinkles
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IncobutolinumtoxinA (Xeomin), 4-injection scheme (Experimental): IncobotulinumtoxinA (Xeomin), also known as 'NT 201' or 'Botulinum toxin type A (150kD), free of complexing proteins' (active ingredient:
  Clostridium Botulinum neurotoxin Type A free of complexing proteins) powder for solution for injection; dose: one injection session of solution, prepared by reconstitution of powder with 0.9% sodium chloride (NaCl); total volume 0.24 mL per side, i.e. 4 x 0.06 mL (4 x 3 units = 12 units); mode of administration: intramuscular injection.
  Interventions: Drug: IncobotulinumtoxinA (Xeomin)
- Placebo 4-injection scheme (Placebo Comparator): Placebo to IncobotulinumtoxinA (Xeomin) powder for solution for injection; dose: one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl; total volume 0.24 mL per side, i.e. 4 x 0.06 mL placebo solution; mode of administration: intramuscular injection.
  Interventions: Drug: Placebo
- IncobotulinumtoxinA (Xeomin), 3-injection scheme (Experimental): IncobotulinumtoxinA (Xeomin), also known as 'NT 201' or 'Botulinum toxin type A (150kD), free of complexing proteins' (active ingredient:
  Clostridium Botulinum neurotoxin Type A free of complexing proteins) powder for solution for injection; dose: one injection session of solution, prepared by reconstitution of powder with 0.9% sodium chloride (NaCl); total volume 0.24 mL per side, i.e. 3 x 0.08 mL (3 x 4 units = 12 units); Mode of administration: intramuscular injection.
  Interventions: Drug: IncobotulinumtoxinA (Xeomin)
- Placebo 3-injection Scheme (Placebo Comparator): Placebo to IncobotulinumtoxinA (Xeomin) powder for solution for injection; dose: one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl; total volume 0.24 mL per side, i.e. 3 x 0.08 mL placebo solution; mode of administration: intramuscular injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IncobotulinumtoxinA (Xeomin) — Intramuscular injection at day 0, at 3 and 4 injection sites per eye (4 x 3 or 3 x 4 units = 12 units per eye)
  Arms: IncobotulinumtoxinA (Xeomin), 3-injection scheme; IncobutolinumtoxinA (Xeomin), 4-injection scheme
Drug: Placebo — Intramuscular injection at day 0, at 3 and 4 injection sites per eye.
  Arms: Placebo 3-injection Scheme; Placebo 4-injection scheme

SUMMARY:
To investigate the efficacy and safety of incobotulinumtoxinA (Xeomin) in comparison to placebo in the treatment of moderate to severe lateral periorbital wrinkles at maximum smile and to compare two different application schemes of Xeomin. Each subject will be treated on the right and left eye area, using the same dose but different application schemes (i.e. 3 or 4 injection sites).

DETAILED DESCRIPTION:
Conducted in Europe

ELIGIBILITY:
Main Inclusion Criteria:

- Moderate (grade 2) to severe (grade 3) symmetrical lateral periorbital wrinkles assessed by the investigator according to the 4-point scale at maximum smile

Main Exclusion Criteria:

- Significant facial asymmetry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Response assessed by an independent rater at maximum smile at week 4 for either eye area compared to baseline. | Week 4
  Responder: subjects with improvement of at least 1 point on a 4 point scale for lateral periorbital wrinkles.

SECONDARY OUTCOMES:
Response assessed by the investigator at maximum smile for either eye area compared to baseline. | Weeks 2, 4, 12, and 20
  Responder: subjects with improvement of at least 1 point on a 4 point scale for lateral periorbital wrinkles.
Response assessed by the subject's global assessment at maximum smile for either eye area compared to baseline. | Weeks 2, 4, 12, and 20
  Responder: subjects with at least a moderate improvement, i.e. a score of at least +2 on a 9 point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: David Eccleston, MD, Principal Investigator — MediZen, Sutton Coldfield, United Kingdom
Locations (12):
- France (3):
  - Cannes
  - Nice
  - Paris
- Germany (4):
  - Düsseldorf
  - Karlsruhe
  - Munich
  - Starnberg
- Roma, Italy
- United Kingdom (4):
  - Bexley. Kent
  - Glasgow
  - London
  - Sutton Coldfield